CLINICAL TRIAL: NCT05871918
Title: A Multicenter, Randomized, Open, Phase III Trial of ddEC-THP（Epirubicin，Cyclophosphamide，TAX(Taxol)，Trastuzumab，Pertuzumab）vs Evaluating the Efficacy and Safety of TCHP （CBP(Carboplatin),TXT(Taxotere),Trastuzumab，Pertuzumab）Neoadjuvant Therapy for HER2-positive Breast Cancer
Brief Title: A Multicenter, Randomized, Open, Phase III Trial of ddEC-THPvs Evaluating the Efficacy and Safety of TCHP Neoadjuvant Therapy for HER2-positive Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIH-TZS-20201008-01
Record Dates: First submitted 2023-05-15; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2022-10

CONDITIONS: HER-2 Positive Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCbHP (Experimental): Experimental group (TCbHP) :
  Taxotere (75mg/m2) + Carboplatin (AUC=5)
  Trastuzumab 6mg/kg(initial dose 8mg/kg)
  Pertuzumab 420mg(initial dose 840mg)
  1/21d times 6 cycle
  Interventions: Drug: TCbHP VS ddEC-THP
- ddEC-THP (Placebo Comparator): Epirubicin (90mg/m2)+ cyclophosphamide (600mg/m2) 1/14d×4 cycle
  Taxol (80mg/m2) 1/7d x 12w
  Trastuzumab 6mg/kg(initial dose 8mg/kg) 1/21d ×4 cycles
  Pertuzumab 420mg(initial dose 840mg) 1/21d x 4 cycles
  Interventions: Drug: TCbHP VS ddEC-THP

INTERVENTIONS:
Drug: TCbHP VS ddEC-THP — The efficacy was evaluated every two cycles, and the effective patients (CR, PR, SD) were treated with surgery after 6 cycles. If treatment does not work, change the treatment plan according to the clinician's decision.

SUMMARY:
The study is being conducted to assess the efficacy and safety of anthracycline-containing ddEC-THP intensive regimen and an anthracycline-free TCbHP neoadjuvant therapy for HER2-positive breast cancer

DETAILED DESCRIPTION:
A Multicenter, Randomized, Open, Phase III，The study is being conducted to assess the efficacy and safety of anthracycline-containing ddEC-THP intensive regimen and an anthracycline-free TCbHP neoadjuvant therapy for HER2-positive breast cancer,Subjects will be treated until disease progression, toxicity is intolerable, informed consent is withdrawn, and investigators determine that medication must be discontinued. Drug efficacy and safety data will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 ~70 years old, female;
2. Histologically confirmed patients with previously untreated stage Ⅱ-Ⅲ HER2-positive breast cancer;
3. HER-2 positive breast cancer, defined as immunohistochemical (IHC) detection of 3+ or in situ hybridization (FISH) results of HER2 gene amplification;
4. There is at least one measurable objective lesion according to RECIST 1.1 criteria;
5. ECOG Physical fitness score is 0-2;
6. Left ventricular ejection fraction LVEF≥50%;
7. Bone marrow function: neutrophils ≥1.5×109/L, platelets ≥100×109/L, hemoglobin ≥90g/L;
8. Liver and kidney function: serum creatinine ≤1.5 times the upper limit of normal value; AST and ALT≤2.5 times the upper limit of normal, or ≤5 times the upper limit of normal in the presence of liver metastasis; Total bilirubin ≤1.5 times the upper limit of normal, or ≤2.5 times the upper limit of normal in patients with Gilbert's syndrome, creatinine clearance greater than 30 mL/min;
9. For female patients who are not menopausal or have not been surgically sterilized: consent to abstinence or use an effective contraceptive method during treatment and for at least 7 months after the last dose in the study treatment
10. The patient has good compliance with the planned treatment, can understand the research process of the study and sign the written informed consent.

Exclusion Criteria:

1. Stage IV (metastatic) breast cancer patients;
2. Patients with inflammatory breast cancer
3. Serious heart disease or discomfort, including but not limited to:

   * History of heart failure or systolic dysfunction (LVEF < 50%)
   * High-risk uncontrolled arrhythmias such as atrial tachycardia, resting heart rate > 100 bpm, significant ventricular arrhythmias (e.g., ventricular tachycardia) or higher-grade atrioventricular block (i.e., Mobitz II second-degree atrioventricular block or third-degree atrioventricular block) Angina pectoris that requires antiangina medication
   * valvular heart disease of clinical significance
   * ECG showed transmural myocardial infarction
   * Poor hypertension control (systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 100 mmHg)
4. Known allergic history of drug components of this protocol; A history of immunodeficiency, including HIV positive, or other acquired, congenital immunodeficiency diseases, or a history of organ transplantation;
5. Patients with severe systemic infection or accompanied by other serious diseases;
6. Have developed other malignant tumors within the previous 5 years, except for cured cervical carcinoma in situ and non-melanoma skin cancer;
7. Pregnant and lactating women, fertile women who tested positive for baseline pregnancy tests, or patients of childbearing age who were unwilling to take effective contraceptive measures during the entire trial period and within 6 months after the last study;
8. Patients who participated in other studies within 30 days prior to the first dose of the investigational drug;
9. Patients deemed unsuitable for this study by the investigator.
10. The patient has good compliance with the planned treatment, can understand the research process of the study and sign the written informed consent.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 832 (Estimated)
Dates: Start 2022-10-08 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
pCR rate using the definition of ypT0/Tis ypN0 (i.e., no invasive residual in breast or nodes; noninvasive breast residuals allowed) at the time of definitive surgery | Up to approximately 24 weeks
  pCR rate (ypT0/is，ypN0) is defined as the percentage of participants without residual invasive tumor on hematoxylin and eosin evaluation of breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy by current AJCC staging criteria assessed by the local pathologist at the time of definitive surgery in all participants.

SECONDARY OUTCOMES:
Event-Free Survival (EFS) | Up to approximately 3 years
  EFS is defined as the time from start of study treatment to any of the following events: progression of disease that precludes surgery, local or distant recurrence, second primary malignancy (breast or other cancers) or death due to any cause.
Invasive Disease-Free Survival (iDFS) | Up to approximately 3 years
  iDFS events are defined as follows: (1)Ipsilateral invasive breast tumor recurrence. (2) Ipsilateral local-regional invasive breast cancer recurrence. (3) Ipsilateral second primary invasive breast cancer. (4) Contralateral invasive breast cancer. (5) Distant recurrence. (6) Death attributable to any cause.
Overall survival (OS) | Up to approximately 3 years
  OS is defined as the time from randomization to death due to any cause. Participants without documented death at the time of the analysis will be censored at the date of the last follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Breast Oncology, Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No